CLINICAL TRIAL: NCT00385138
Title: A Clinical Trial Comparing Treatment With Cangrelor (in Combination With Usual Care) to Usual Care, in Subjects Who Require Percutaneous Coronary Intervention (PCI).
Brief Title: Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition.
Acronym: Platform
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient evidence of the clinical effectiveness of cangrelor
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMC-CAN-05-03
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Atherosclerosis; Acute Coronary Syndrome (ACS)
Keywords: Percutaneous Coronary Intervention (PCI); ACS
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome | interventions — cangrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cangrelor (Experimental): cangrelor bolus (30 mcg/kg) & infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion) + placebo capsules (to match) at end of PCI + active clopidogrel (600mg) immediately post infusion
  Interventions: Drug: Cangrelor; Drug: clopidogrel; Drug: Placebo capsules - end of PCI
- Clopidogrel (Active Comparator): placebo bolus & infusion (to match) + clopidogrel capsules (600 mg) at end of PCI + placebo capsules (to match) immediately post infusion
  Interventions: Drug: clopidogrel; Drug: Placebo bolus & placebo infusion; Drug: Placebo capsules - end of infusion

INTERVENTIONS:
Drug: Cangrelor — cangrelor bolus (30 mcg/kg) & cangrelor infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion)
  Arms: Cangrelor
Drug: clopidogrel — clopidogrel capsules (600 mg) at end of PCI
  Other Names: Plavix
Drug: Placebo bolus & placebo infusion — placebo bolus (30 mcg/kg) & placebo infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion)
  Arms: Clopidogrel
Drug: Placebo capsules - end of PCI — Placebo capsules given at the end of PCI to mimic 600mg clopidogrel dosing
  Arms: Cangrelor
Drug: Placebo capsules - end of infusion — Placebo capsules given at the end of infusion to mimic 600mg clopidogrel dosing
  Arms: Clopidogrel

SUMMARY:
The primary objective of this study is to demonstrate that the efficacy of cangrelor (combined with usual care) is superior to that of usual care, in subjects requiring percutaneous coronary intervention (PCI) as measured by a composite of all-cause mortality, myocardial infarction (MI), and ischemia-driven revascularization (IDR).

ELIGIBILITY:
Inclusion Criteria:

Angiography demonstrating atherosclerosis amenable to treatment by percutaneous coronary intervention (PCI) with or without stent implantation and diagnosis of Acute Coronary Syndrome (ACS) by elevated cardiac markers or ischemic chest discomfort w/electrocardiogram changes + age > 65 or diabetes.

Exclusion Criteria:

1. Not a candidate for PCI
2. ST-segment elevation myocardial infarction (STEMI) within 48 hours of randomization
3. Increased bleeding risk: ischemic stroke within the last year or any previous hemorrhagic stroke, intra-cranial tumor, cerebral arteriovenous malformation, or intracranial aneurysm; recent (<1 month) trauma or major surgery [including coronary artery bypass graft (CABG) surgery]; currently receiving warfarin, active bleeding
4. Impaired hemostasis: known International Normalized Ratio (INR) >1.5 at screening; past or present bleeding disorder (including congenital bleeding disorders such as von Willebrand's disease or hemophilia, acquired bleeding disorders, and unexplained clinically significant bleeding disorders), thrombocytopenia (platelet count <100,000/µL) at screening
5. Severe hypertension not adequately controlled by antihypertensive therapy at the time of randomization
6. Receipt of fibrinolytic therapy in the 12 hours preceding randomization
7. Receipt of any thienopyridine (clopidogrel or ticlopidine) in the 7 days preceding randomization
8. Glycoprotein IIb/IIIa (GPI) Inhibitor usage within the previous 12 hours [applicable to unstable angina (UA) and non-ST-elevation myocardial infarction (NSTEMI) patients]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5364 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simona Skerjanec, PharmD, Study Director — The Medicines Company; Deepak L. Bhatt, MD, Principal Investigator — The Cleveland Clinic; Robert A. Harrington, MD, Principal Investigator — Duke University
Locations (1):
- Innovis Health, Fargo, North Dakota, United States

REFERENCES:
- [Result] Bhatt DL, Lincoff AM, Gibson CM, Stone GW, McNulty S, Montalescot G, Kleiman NS, Goodman SG, White HD, Mahaffey KW, Pollack CV Jr, Manoukian SV, Widimsky P, Chew DP, Cura F, Manukov I, Tousek F, Jafar MZ, Arneja J, Skerjanec S, Harrington RA; CHAMPION PLATFORM Investigators. Intravenous platelet blockade with cangrelor during PCI. N Engl J Med. 2009 Dec 10;361(24):2330-41. doi: 10.1056/NEJMoa0908629. PMID 19915222
- [Derived] Gutierrez JA, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL; CHAMPION Investigators. Efficacy and safety of cangrelor in patients with peripheral artery disease undergoing percutaneous coronary intervention - Insights from the CHAMPION program. Am Heart J Plus. 2021 Aug 25;9:100043. doi: 10.1016/j.ahjo.2021.100043. eCollection 2021 Sep. PMID 38551015
- [Derived] Peterson BE, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL. Effect of Platelet Inhibition by Cangrelor Among Obese Patients Undergoing Coronary Stenting: Insights From CHAMPION. Circ Cardiovasc Interv. 2022 Mar;15(3):e011069. doi: 10.1161/CIRCINTERVENTIONS.121.011069. Epub 2022 Feb 24. PMID 35196863
- [Derived] Groves EM, Bhatt DL, Steg PG, Deliargyris EN, Stone GW, Gibson CM, Hamm CW, Mahaffey KW, White HD, Angiolillo DJ, Prats J, Harrington RA, Price MJ. Incidence, Predictors, and Outcomes of Acquired Thrombocytopenia After Percutaneous Coronary Intervention: A Pooled, Patient-Level Analysis of the CHAMPION Trials (Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition). Circ Cardiovasc Interv. 2018 Apr;11(4):e005635. doi: 10.1161/CIRCINTERVENTIONS.117.005635. PMID 29632238
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Steg G, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Deliargyris EN, Prats J, Mahaffey KW, White HD, Bhatt DL. Short- and long-term mortality following bleeding events in patients undergoing percutaneous coronary intervention: insights from four validated bleeding scales in the CHAMPION trials. EuroIntervention. 2018 Feb 2;13(15):e1841-e1849. doi: 10.4244/EIJ-D-17-00723. PMID 28988157
- [Derived] Parker WA, Bhatt DL, Prats J, Day JRS, Steg PG, Stone GW, Hamm CW, Mahaffey KW, Price MJ, Gibson CM, White HD, Storey RF; CHAMPION PHOENIX Investigators. Characteristics of dyspnoea and associated clinical outcomes in the CHAMPION PHOENIX study. Thromb Haemost. 2017 Jun 2;117(6):1093-1100. doi: 10.1160/TH16-12-0958. Epub 2017 Apr 6. PMID 28382371
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Deliargyris EN, Steg PG, Gibson CM, Hamm CW, Price MJ, Menozzi A, Prats J, Elkin S, Mahaffey KW, White HD, Bhatt DL. Evaluation of Ischemic and Bleeding Risks Associated With 2 Parenteral Antiplatelet Strategies Comparing Cangrelor With Glycoprotein IIb/IIIa Inhibitors: An Exploratory Analysis From the CHAMPION Trials. JAMA Cardiol. 2017 Feb 1;2(2):127-135. doi: 10.1001/jamacardio.2016.4556. PMID 27902833
- [Derived] White HD, Chew DP, Dauerman HL, Mahaffey KW, Gibson CM, Stone GW, Gruberg L, Harrington RA, Bhatt DL. Reduced immediate ischemic events with cangrelor in PCI: a pooled analysis of the CHAMPION trials using the universal definition of myocardial infarction. Am Heart J. 2012 Feb;163(2):182-90.e4. doi: 10.1016/j.ahj.2011.11.001. PMID 22305835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for randomization based on the need for percutaneous coronary intervention (PCI).
  Randomization could only occur after the need for PCI was confirm by angiography.
Period: Overall Study
Arm/Group | Cangrelor | Clopidogrel
Started | 2695 | 2669
Intent-to-treat (ITT) | 2693 (All patients randomized excluding two (2) who withdrew consent for using study data.) | 2669
Modified Intent-to-treat (mITT) | 2656 (Excludes 37 patients who either did not receive study drug or have PCI.) | 2645 (Excludes 24 patients who either did not received study drug or have PCI.)
Safety Population | 2662 (Includes all randomized patients who received at least one dose of study drug.) | 2650 (Includes all randomized patients who received at least one dose of study drug.)
Completed | 2665 ("Completed" means patient completed scheduled visits or developed a primary endpoint event.) | 2641 ("Completed" means patient completed scheduled visits or developed a primary endpoint event.)
Not Completed | 30 | 28

BASELINE CHARACTERISTICS:
Population: mITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cangrelor | Clopidogrel | Total
Number analyzed (Participants) | 2656 | 2645 | 5301
Age, Continuous [Mean (Standard Deviation); unit: years] — mITT population
  years | 62.5 (11.4) | 62.5 (11.3) | 62.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — mITT population
  Participants
    Female | 747 | 782 | 1529
    Male | 1909 | 1863 | 3772
Region of Enrollment [Number; unit: participants] — The analysis by region was performed on the mITT population.
  participants
    United States | 815 | 809 | 1624
    Argentina | 39 | 42 | 81
    Brazil | 48 | 49 | 97
    Bulgaria | 403 | 394 | 797
    Canada | 3 | 2 | 5
    Czech Republic | 342 | 345 | 687
    Georgia | 47 | 43 | 90
    India | 235 | 236 | 471
    Lithuania | 54 | 55 | 109
    New Zealand | 22 | 20 | 42
    Belarus | 33 | 31 | 64
    Russian Federation | 215 | 218 | 433
    Slovakia | 33 | 27 | 60
    South Africa | 102 | 100 | 202
    Korea, Republic of | 159 | 166 | 325
    Spain | 17 | 21 | 38
    Thailand | 58 | 58 | 116
    Netherlands | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All-cause Mortality, Myocardial Infarction (MI), and Ischemia-driven Revascularization (IDR)
Description: mITT population; (composite incidence)
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 185 | 210

2. Secondary Outcome: Incidence of All-cause Mortality or MI
Description: mITT population
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 180 | 204

3. Secondary Outcome: Incidence of All-cause Mortality
Description: mITT population
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 6 | 18

4. Secondary Outcome: Incidence of MI
Description: mITT population
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 177 | 191

5. Secondary Outcome: Incidence of IDR
Description: mITT population
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 19 | 24

6. Secondary Outcome: Incidence of Stent Thrombosis
Description: mITT population
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 5 | 16

7. Secondary Outcome: Incidence of Stroke
Description: mITT
Time Frame: randomization through 48 hours post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2654 | 2641
participants | 7 | 5

8. Secondary Outcome: Incidence of All-cause Mortality
Description: mITT population
Time Frame: randomization through 1 year post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2628 | 2618
participants | 94 | 113

9. Secondary Outcome: Incidence of Procedure Events [Abrupt Closure, Threatened Abrupt Closure, Need for Urgent Coronary Artery Bypass Graft (CABG) Surgery, Unsuccessful Procedure, New Thrombus or Suspected Thrombus, and/or Acute Stent Thrombosis]
Description: mITT population A patient could have multiple procedural events.
Time Frame: During index PCI
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2656 | 2645
participants | 122 | 142

10. Secondary Outcome: Incidence of GUSTO Severe / Life-threatening
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours post randomization
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2662 | 2650
participants | 9 | 6

11. Secondary Outcome: Incidence of Thrombolysis in Myocardial Infarction (TIMI) Major
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours post randomization
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2662 | 2650
participants | 4 | 9

12. Secondary Outcome: Incidence of ACUITY Major Bleeding
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours post randomization
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2662 | 2650
participants | 145 | 91

13. Secondary Outcome: Incidence of ACUITY Major Bleeding Without Hematoma >/= 5 cm
Description: Major bleeding (non-CABG-related) - Safety population excludes ACUITY major bleeding for which the only qualifying event was hematoma >/= 5 cm.
Time Frame: randomization through 48 hours post randomization
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2662 | 2650
participants | 43 | 29

14. Secondary Outcome: Incidence of All-cause Mortality, MI, or IDR
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 227 | 249

15. Secondary Outcome: Incidence of All-cause Mortality or MI
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 213 | 233

16. Secondary Outcome: Incidence of All-cause Mortality
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 35 | 45

17. Secondary Outcome: Incidence of MI
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 189 | 201

18. Secondary Outcome: Incidence of IDR
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 37 | 46

19. Secondary Outcome: Incidence of Stent Thrombosis
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 15 | 28

20. Secondary Outcome: Incidence of Stroke
Description: mITT population
Time Frame: randomization through 30 days post randomization
Population: mITT population, based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor | Clopidogrel
Number analyzed (Participants) | 2647 | 2629
participants | 6 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 48 hours after study drug initiation
Description: The analysis population used for adverse event reporting is the Safety Population.
Arm/Group | Cangrelor | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 48/2662 | 55/2650
Other Adverse Events (participants affected / at risk) | 596/2662 | 530/2650
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cangrelor (N=2662) | Clopidogrel (N=2650)
atrial fibrillation (Cardiac disorders) | 2 | 1
atrioventricular block (Cardiac disorders) | 0 | 1
cardiac arrest (Cardiac disorders) | 1 | 3
cardiac failure acute (Cardiac disorders) | 1 | 0
cardiac failure congestive (Cardiac disorders) | 3 | 1
cardiac tamponade (Cardiac disorders) | 0 | 1
cardiogenic shock (Cardiac disorders) | 6 | 11
coronary artery dissection (Cardiac disorders) | 0 | 2
coronary artery occlusion (Cardiac disorders) | 0 | 1
coronary artery perforation (Cardiac disorders) | 1 | 0
coronary artery thrombosis (Cardiac disorders) | 0 | 1
electromechanical dissociation (Cardiac disorders) | 1 | 3
ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
left ventricular failure (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 0
myocardial rupture (Cardiac disorders) | 0 | 1
pericardial effusion (Cardiac disorders) | 1 | 0
sick sinus syndrome (Cardiac disorders) | 1 | 0
torsade de pointes (Cardiac disorders) | 0 | 2
ventricular arrhythmia (Cardiac disorders) | 1 | 0
ventricular fibrillation (Cardiac disorders) | 4 | 2
ventricular tachycardia (Cardiac disorders) | 1 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
chest discomfort (General disorders) | 1 | 1
chest pain (General disorders) | 2 | 1
non-cardiac chest pain (General disorders) | 1 | 0
pyrexia (General disorders) | 2 | 0
bacterial sepsis (Infections and infestations) | 0 | 1
lung infection (Infections and infestations) | 0 | 1
arterial injury (Injury, poisoning and procedural complications) | 0 | 1
brain contusion (Injury, poisoning and procedural complications) | 1 | 0
head injury (Injury, poisoning and procedural complications) | 1 | 0
thrombosis in device (Injury, poisoning and procedural complications) | 0 | 2
anticoagulation drug level below therapeutic (Investigations) | 1 | 0
cardiac enzymes increased (Investigations) | 1 | 0
troponin increased (Investigations) | 0 | 1
dizziness (Nervous system disorders) | 1 | 0
dizziness postural (Nervous system disorders) | 0 | 1
haemorrhage intracranial (Nervous system disorders) | 1 | 0
migraine (Nervous system disorders) | 1 | 0
myelitis (Nervous system disorders) | 0 | 1
transient ischaemic attack (Nervous system disorders) | 0 | 2
nephropathy toxic (Renal and urinary disorders) | 2 | 0
renal failure chronic (Renal and urinary disorders) | 1 | 0
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0
hypertension (Vascular disorders) | 1 | 2
hypertensive emergency (Vascular disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 4
peripheral ischaemia (Vascular disorders) | 0 | 1
vascular pseudoaneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cangrelor (N=2662) | Clopidogrel (N=2650)
back pain (Musculoskeletal and connective tissue disorders) | 91 | 85
chest pain (General disorders) | 73 | 69
nausea (Gastrointestinal disorders) | 71 | 66
headache (Nervous system disorders) | 60 | 68
hypotension (Vascular disorders) | 43 | 38
dyspnea (Respiratory, thoracic and mediastinal disorders) | 38 | 15
vomiting (Gastrointestinal disorders) | 37 | 31
pyrexia (General disorders) | 36 | 20
hypertension (Vascular disorders) | 28 | 22
puncture site pain (General disorders) | 21 | 29
pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 14
pain (General disorders) | 14 | 8
chest discomfort (General disorders) | 13 | 11
syncope vasovagal (Nervous system disorders) | 13 | 4
anxiety (Psychiatric disorders) | 13 | 3
angina pectoris (Cardiac disorders) | 11 | 17
bradycardia (Cardiac disorders) | 10 | 15
insomnia (Psychiatric disorders) | 10 | 15

LIMITATIONS AND CAVEATS:
Discontinued per prespecified stopping rules after the 70% interim analyses was conducted indicating the trial was not likely not meet the goal of demonstrating superiority to clopidogrel administered as usual care. No safety issues were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI communications regarding trial results are prohibited until after the communication and publication of the multi-center results by Sponsor, but no more than 12 months after conclusion of the trial at all sites.

PI must submit results communications to sponsor for review at least 40 days prior to submission for publication and Sponsor may embargo such communications for a period that is less than or equal to 135 days solely to seek appropriate patent protection.